CLINICAL TRIAL: NCT03367481
Title: Evaluation of Gingival Fissures Associated With Soft and Medium Toothbrushes: Crossover Randomized Clinical Trial
Brief Title: Evaluation of Gingival Fissures Associated With Soft and Medium Toothbrushes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Rui Vicente Oppermann, Head Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Gingival fissures study
Record Dates: First submitted 2017-12-01; First posted 2017-12-08 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Gingival Recession; Gingival Abrasion; Wounds and Injuries
Keywords: Gingival fissures; Gingival recession; Risk factors; Traumatic toothbrushing
MeSH Terms: conditions — Gingival Recession; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control toothbrush (Active Comparator): The participants will use a toothbrush with soft bristles.
  Interventions: Device: Toothbrush type
- Test toothbrush (Experimental): The participants will use a toothbrush with medium bristles.
  Interventions: Device: Toothbrush type

INTERVENTIONS:
Device: Toothbrush type — In this cross-over study, the participants will use either a soft brush (control) and the medium brush (test).

SUMMARY:
Gingival fissures (GF) have been suggested as risk indicators for clinical attachment loss (CAL) and gingival recession, especially in free surfaces and in patients with low plaque scores. The major factors related to the GF occurrence are high daily brushing frequencies, excessive force to brush, malpositioned teeth, use of abrasive dentifrices, and stiffness of the toothbrushes bristles. Thus, in order to better understand the pathogenesis and progression of GF, this study aim to evaluate the incidence and behavior of GF in young adults using soft and medium brushes, in a cross-over randomized clinical trial along 6 months.

DETAILED DESCRIPTION:
Material and Methods: A blinded crossover randomized clinical trial will be conducted with 20 patients from a school (Colégio Tiradentes da Brigada Militar) at Porto Alegre city, southern of Brazil. Patients, aged between 18 to 25 years old, having at least 20 teeth, without previous history of periodontitis [clinical attachment loss (CAL) ≥ 3mm], and good systemic health will be included if they do not have orthodontic appliances or dental implants, or dental caries or restorations at cervical surface. Data collection will performed by two trained, calibrated and blinded examiners, and will comprehend a brief interview regarding oral hygiene and deleterious habits, full-mouth exams (6 sites/tooth) of Plaque Index (PlI), Gingival Index (GI), Pocket Probing Depth (PPD), and CAL, and clinical photographs (from 1st and 2nd premolars and 1st molar area in all quadrants) under disclosing solution (2Tone®) to evaluate the presence of gingival fissures (GF). After baseline data collection the participants will be randomized in one of the experimental groups according the toothbrush bristles stiffness: G1) soft; or G2) medium. No oral hygiene instruction will be provided to groups, and the patients will not be informed about the type of brush that will be provided. Re-exams (PlI, GI and photographs) will be conducted at 30, 60, 90 days. At day 90 the 1st phase will be finished, and the participants will have a 10-days wash-out period. At day 100, the 2nd phase will start, and the participants will change the groups. Re-exams will be conducted at 130, 160, 190 days. At day 190, the study will be finished. The participants will be oriented to return the toothbrushes used at the end of each experimental phase.

Outcomes: The primary outcome will be the number of participants with GF observed over the study period. Also, the incidence, size and duration of the GF will be compared regarding the variables: type of bristle, self-reported toothbrushing frequency, toothbrush deformation, and deleterious habits. McNemar test will be used to compare the frequencies of patients with GF and the number of lesions observed both inter and intra-groups. Uni- and multivariate regression models will be conducted to determine associations between the outcome and independent variables. The mean number of new fissures, GF that decreased, and GF that stabilized over time will be compared inter-groups as secondary analysis. Intention-to-treat analysis will be conducted, considering the individual the unit of analysis and a α-error of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* have at least 20 teeth,
* negative history of periodontitis (CAL ≥ 3mm),
* good systemic health.

Exclusion Criteria:

* do not have orthodontic appliances or dental implants,
* absence of dental caries or restorations at cervical buccal surface.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Gingival fissures associated with toothbrushing | 6 months
  Standardized photographs, under disclosing solution (2Tone®) from 1st and 2nd premolars and 1st molar area in all quadrants, will be taken at baseline and at days 30, 60, 90, 100, 130, 160 and 190 for evaluation of gingival fissures. The disclosing solution is safe, without contra-indications in the literature and facilitates visualization of gingival lesions and plaque. After, the photographs will be analyzed in an image software in order to determine the mean number of new fissures, fissures that decreased, and those that stabilized over time. If, at any time during the study a gingival fissure become greater than 3mm, the patients will stop the use of the specific toothbrush and will be follow until the regression of the lesion.

SECONDARY OUTCOMES:
Toothbrush wear | 6 months
  The participants will be oriented to return the toothbrushes used at the end of each experimental phase. The toothbrush deformation/wear will be investigated by comparing the dimensions of height, width and length, in anterior, middle and posterior parts of the toothbrush (measured with a digital caliper), before and after its use by the participants, in each phase of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Rui V Oppermann, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil